CLINICAL TRIAL: NCT07011108
Title: Machine Learning for Estimating Cardiorespiratory Fitness in Patients With Obesity
Acronym: FitML-O
Status: Active, not recruiting | Type: Observational
Sponsor: Sykehuset i Vestfold HF (Other)
Responsible Party: Principal Investigator, Jarle Berge, Phd, associate professor, Sykehuset i Vestfold HF
Other Study IDs: FitML-O
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Obesity; Overweight
Keywords: Obesity; overweight; Cardiorespiratory fitness; VO2max; Machine learning; ML, web-application;
MeSH Terms: conditions — Obesity; Overweight | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention (observational study) — no intervention

SUMMARY:
The primary aim of this study is to develop an obesity-specific machine learning (ML) model capable of accurately estimating VO2max, a key indicator of cardiovascular fitness.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with severe obesity
* body mass index (BMI) ≥40.0 kg •m-2, or 35.0-39.9 kg •m-2 with at least one obesity-related comorbidity

Exclusion Criteria:

* not obese

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with obesity from Norway
Sampling Method: Non-Probability Sample
Enrollment: 1700 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2027-12-10 (Estimated); Study Completion 2027-12-24 (Estimated)

PRIMARY OUTCOMES:
Machine learning model to estimate vo2max | The project will be completed in 2027
  The primary aim of this study is to develop an obesity-specific ML model capable of accurately estimating VO2max, a key indicator of cardiovascular fitness

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to confidentiality concerns, lack of participant consent for data sharing, or institutional policy restrictions.